CLINICAL TRIAL: NCT04734262
Title: A Phase II Study to Explore the Safety, Tolerability, and Preliminary Antitumor Activity of Sitravatinib Plus Tislelizumab or Combination With Nab-paclitaxel in Patients With Locally Recurrent or Metastatic Triple Negative Breast Cancer (TNBC)
Acronym: SPARK
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Chief Physician, Fudan University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-900-2001-IIT
Record Dates: First submitted 2021-01-29; First posted 2021-02-02 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — sitravatinib; tislelizumab; 130-nm albumin-bound paclitaxel; Taxes

STUDY DESIGN:
Intervention Model Description: Cohort A Subjects will receive 70mg sitravatinib in combination with 200mg tislelizumab until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Cohort B Subjects will receive 100mg sitravatinib in combination with 200mg tislelizumab until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Cohort C Subjects will receive sitravatinib in combination with 200mg tislelizumab and 100 mg/m2 nab-paclitaxel until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
Masking Description: None (Open Label)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Subjects will receive 70mg sitravatinib in combination with 200mg tislelizumab until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Sitravatinib; Drug: Tislelizumab
- Cohort B (Experimental): Subjects will receive 100mg sitravatinib in combination with 200mg tislelizumab until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Sitravatinib; Drug: Tislelizumab
- Cohort C (Experimental): Subjects will receive sitravatinib in combination with 200mg tislelizumab and 100 mg/m2 nab-paclitaxel until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Sitravatinib; Drug: Tislelizumab; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Sitravatinib — Sitravatinib QD PO Sitravatinib is a small molecule inhibitor of receptor tyrosine kinases
  Other Names: MGCD516
Drug: Tislelizumab — Tislelizumab Q3W IV Tislelizumab is a programmed death receptor-1 (PD-1) blocking antibody
  Other Names: BGB-A317
Drug: Nab-paclitaxel — Nab-paclitaxel D1, D8 Q3W IV Nab-paclitaxel is a chemotherapy drug which combines the chemotherapy drug paclitaxel with albumin
  Other Names: Nanoparticle albumin-bound paclitaxel
  Arms: Cohort C

SUMMARY:
The purpose of this study is to assess the efficacy and safety of sitravatinib plus tislelizumab or combination with nab-paclitaxel in locally recurrent or metastatic triple-negative breast cancer (TNBC) patients.

DETAILED DESCRIPTION:
This is a prospective, single-center, three cohorts, phase II clinical trial in locally recurrent or metastatic triple-negative breast cancer(TNBC) patients. Subjects will be divided into three cohorts by different treatment combination. Cohort A & Cohort B aim to explore the two dosages of sitravatinib in combination with tislelizumab in TNBC with prior ≤ 3 treatment line. Cohort A patients will receive 70mg sitravatinib (QD PO) in combination with 200mg tislelizumab (Q3W IV); Cohort B patients will receive 100mg sitravatinib (QD PO) in combination with 200mg tislelizumab (Q3W IV). Cohort C aims to explore the sitravatinib (QD PO) plus 200mg tislelizumab (Q3W IV) and 100 mg/m2 nab-paclitaxel (D1, D8 Q3W IV) in TNBC previously untreated for metastatic setting or recurred/metastasized after surgery. Subjects in the three cohorts will be treated until disease progression, intolerable toxicity, informed consent withdrawn, or investigators-determined medication termination. Drug efficacy and safety data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments
* Age ≥ 18 years on the day of signing the ICF (or the legal age of consent in the jurisdiction in which the study is taking place)
* Histologically confirmed diagnosis of TNBC characterized by estrogen-receptor negative (ER-), progesterone receptor negative (PR-) and human epidermal growth factor-2 receptor negative (HER2-);
* ≤ 3 prior lines of systemic therapy
* For patients refractory/resistant to anti-PD-1/PD-L1 antibodies, there should be no anti-PD-1/PD-L1 treatment-related toxicity from prior therapies
* Previously untreated for metastatic setting or recurred/metastasized after surgery for locally recurrent or metastatic breast cancer (cohort C), and the time from previous neo-/adjuvant therapy to recurrence met the following requirements: ≥ 6 months interval between the end of neo-/adjuvant paclitaxel-based treatment and the onset of recurrence/metastasis; ≥ 6 months interval between the end of neo-/adjuvant anti-angiogenic treatment and the onset of recurrence/metastasis; ≥ 6 months interval between the end of neo-/adjuvant immunotherapy and recurrence/metastasis
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function
* Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and ≥ 120 days after the last dose of study drug(s), and have a negative serum pregnancy test ≤ 7 days of first dose of study drug(s)
* Nonsterile males must be willing to use a highly effective method of birth control for the duration of the study and for ≥ 120 days after the last dose of study drug(s)

Exclusion Criteria:

* Active leptomeningeal disease or uncontrolled brain metastasis
* Active autoimmune diseases or history of autoimmune diseases that may relapse
* Any active malignancy ≤ 2 years
* Severe chronic or active infections (including tuberculosis infection, etc) requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days prior to first dose of study drug(s)
* History of interstitial lung disease, noninfectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases, etc
* Known history of human immunodeficiency virus (HIV) infection
* Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers
* Any major surgical procedure requiring general anesthesia ≤ 28 days before the first dose of study drug(s)
* Prior allogeneic stem cell transplantation or organ transplantation
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Bleeding or thrombotic disorders or use of anticoagulants such as warfarin or similar agents requiring therapeutic international normalized ratio (INR) monitoring
* Any systemic chemotherapy within 28 days of the first dose of study drug(s) or hormone therapy, targeted therapy, or any investigational therapies Toxicities (as a result of prior anticancer therapy) that have not recovered to baseline or stabilized, except for AEs not considered a likely safety risk (eg, alopecia, neuropathy, and specific laboratory abnormalities)
* Inability to swallow capsules or disease significantly affecting gastrointestinal function
* Pregnant or breastfeeding woman NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) by Investigator in Cohort A, Cohort B and Cohort C | Up to 12 months
  The number of people with tumor responses according to RECIST (V1.1): the proportion of participants who achieves a best overall response of complete response (CR) or partial response (PR).
Number of participants experiencing ≥ Grade 3 TRAEs in Cohort B | Up to 12 months
  TRAE are adverse events that occur during or after the first administration of the study drug until 30 days after the study drug is discontinued or the new anticancer treatment is initiated.

SECONDARY OUTCOMES:
Duration of Response (DOR) by Investigator in Cohort A, Cohort B and Cohort C | Up to 12 months
  The time from the date that response criteria are first met to the date that progressive disease (PD) is objectively documented or death, whichever occurs first.
Disease Control Rate (DCR) by Investigator in Cohort A, Cohort B and Cohort C | Up to 12 months
  The proportion of participants who achieves a best overall response of CR, PR or stable disease(SD).
Progression-free Survival (PFS) by Investigator in Cohort A, Cohort B and Cohort C | Up to 12 months
  Time from the date of randomization to the date of progressive disease (PD) or death, whichever occurs first.
One-year overall survival (OS) rate in Cohort A, Cohort B and Cohort C | Up to 12 months
  OS defined as the time from the date of randomization to the date of death due to any reason. One-year survival rate (percentage of subjects alive at 1 year) was estimated from OS data.
Number of participants experiencing Adverse Events (AEs), Treatment-Related Adverse Events (TRAEs) or Serious Adverse Events (SAEs) in Cohort A, Cohort B and Cohort C | Up to 12 months
  Adverse Events (AEs) according to CTCAE v5.0
Patient report outcomes (PROs) based on the EORTC QLQ-C30 (V.3) Quality of Life Questionnaire in Cohort B and Cohort C | Through study completion, an average of 1 year
  Evaluating the Quality of Life of participants as assessed by EORTC QLQ-C30 Questionnaire
Potential biomarkers associated with efficacy, drug resistance, and/or disease progression (PD) in tumor tissues in Cohort A, Cohort B and Cohort C | Through study completion, an average of 1 year
  Potential biomarkers in tumor tissues associated with efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Lei Fan, Xiyu Liu, Xi Jin, Yunsong Yang, Li Chen, Xin Hu, Zhonghua Wang, Yizhou Jiang, and Zhimin Shao. The safety, tolerability, and preliminary antitumor activity of sitravatinib plus tislelizumab in patients with locally recurrent or metastatic triple-negative breast cancer.Journal of Clinical Oncology 2022 40:16_suppl, 1070-1070
- [Result] L. Liu, X. Jin, Y. Xu, S. Wu, Y. Yang, L. Chen, W. Zhang, L. Ma, X. Hu, Z. Wang, Y. Jiang, Z. Shao. The safety, tolerability, and preliminary antitumor activity of sitravatinib plus tislelizumab in patients (pts) with locally recurrent or metastatic triple negative breast cancer (TNBC): a multi-cohort, phase II trial. Annals of Oncology (2022) 16 (suppl_1): 100102-100102. 10.1016/iotech/iotech100102